CLINICAL TRIAL: NCT05402423
Title: An Integrated Intervention of Computerized Cognitive Training and Physical Exercise in Virtual Reality for People With Alzheimer's Disease: the JDome Study Protocol
Brief Title: An Integrated Intervention of Computerized Cognitive Training and Physical Exercise in Virtual Reality for People With Alzheimer's Disease (JDome)
Acronym: JDome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not possible to acquire the medical device
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Fondazione Cariverona, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INRCA_003_2022
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; virtual system; aerobic exercise; cognitive training; dementia; quality of life
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JDome rehabilitation group (Experimental): Patients will undergo cognitive training with Brainer web platform via tablet followed by aerobic exercise with the JDome System
  Interventions: Device: Computerized cognitive training plus aerobic exercise with the JDome System
- control group (Active Comparator): Patients will undergo cognitive training with Brainer web platform via tablet followed by aerobic exercise with standard exercise bike
  Interventions: Device: Computerized cognitive training plus aerobic exercise with standard exercise bike

INTERVENTIONS:
Device: Computerized cognitive training plus aerobic exercise with the JDome System — Sixteen treatment sessions of 60 minutes will be conducted (2 training sessions per week, for 8 weeks).
  Each session will involve the following activities:
  * 30 minutes of computerized cognitive training with the Brainer web platform, a medical device that contains 78 exercises in the five cognitive areas involved in the degeneration process of dementia
  * 30 minutes of aerobic training with the JDOME system,
  Arms: JDome rehabilitation group
Device: Computerized cognitive training plus aerobic exercise with standard exercise bike — Sixteen treatment sessions of 60 minutes will be conducted (2 training sessions per week, for 8 weeks).
  Each session will involve the following activities:
  * 30 minutes of computerized cognitive training with the Brainer web platform, a medical device that contains 78 exercises in the five cognitive areas involved in the degeneration process of dementia
  * 30 minutes of aerobic training with standard exercise bike
  Arms: control group

SUMMARY:
JDOME is a randomized controlled trial to test the effectiveness of a computerized cognitive training with the Brainer web platform and aerobic training with the JDOME system vs. a computerized cognitive training with the Brainer web platform and aerobic training with a standard exercise bike in subjects with Alzheimer's Disease at early stage. The JDome BikeAround is a tool that take people with dementia on a virtual bicycle tour along the paths of memories. It combines an exercise bike, a dome-shaped projector and Google Street View technology.

DETAILED DESCRIPTION:
JDOME study is designed as a randomized controlled trial to test the effectiveness of a training that combines the JDome virtual reality system for aerobic exercise with computerized cognitive training via tablet. The Experimental Group (EG) will receive computerized cognitive training with the Brainer web platform and aerobic training with the JDOME system (a tool that combines an exercise bike, a dome-shaped projector and Google Street View technology).The Control Group (CG) will receive computerized cognitive training with the Brainer web platform and aerobic training with a standard exercise bike.

Assessment will be performed at the baseline (T0), at the end of intervention (after eight weeks -T1) and 12 weeks after the end of intervention (follow-up T2).

The primary aim is to assess the stabilization of the global cognition of people with mild-stage Alzheimer's disease at the Mini-Mental State Examination (MMSE) and at the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog); The secondary aim is the analyses of the modification of the quality of life, mood, behavioral disturbances, and physical function in people with mild-stage Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and over;
* Pre-existing diagnosis of Alzheimer's, in mild phase, according to the 2011 criteria of the National Institute on Aging-Alzheimer's Association (NIA-AA);
* Clinical Dementia Rating Scale CDR = 1;
* Mini Mental State Examination MMSE > 19;
* Functional Ambulation Categories FAC ≥4;
* Tinetti scale ≥ 20;
* Presence of a contact family caregiver
* Reside at home

Exclusion Criteria:

* Failure to meet the inclusion criteria
* Sensory deficits not compensated by the use of prostheses
* Psychological and behavioral disorders not compensated by drug treatment
* Medical contraindication to moderate intensity aerobic exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-27 (Estimated); Primary Completion 2023-06-26 (Estimated); Study Completion 2023-06-26 (Estimated)

PRIMARY OUTCOMES:
change in cognitive impairment | baseline, 8, and 22 weeks later
  Mini-Mental State Examination was designed as a clinical method for grading cognitive impairment. The score ranges from 0 to 30: scores ≥ 24 indicate normality, between 18-23 indicate mild cognitive impairment, between 11-17 moderate cognitive deficits, scores ≤ 10 severe cognitive impairments. The reported score will be corrected according to age and education.
change in short and medium term memory | baseline, 8 and 22 weeks later
  Alzheimer's Disease Assessment Scale (ADAS-cog) consists of 11 items that investigate: short and medium term memory, language, praxia (simple, constructive, ideational), temporal-spatial orientation. The score ranges from 0 (no cognitive impairment) to 70 (maximum cognitive impairment).

SECONDARY OUTCOMES:
change in quality of life | baseline and 8, 22 weeks later
  Alzheimer's Disease scale (QoL-AD) includes 13 items that evaluate subjective (eg, perceived quality of life and psychological well-being) and objective (eg, behavioral competence and environment) components of the quality of life. Items are rated by subjects with dementia on a 4-point scale from 1 (poor) to 4 (excellent). Higher scores indicate a better quality of life.
change in physical performance | baseline, 8 and 22 weeks later
  Short Physical Performance Battery (SPPB) is a short battery of tests designed to assess the function of the lower limbs. This scale consists of 3 different sections: balance assessment, evaluation of walking on 4 linear meters, evaluation of the ability to perform, for 5 consecutive times, the sit to stand from a chair, without using the upper limbs. The total scale score therefore has a range from 0 to 12. A total score below 10 indicates frailty and a high risk of disability and falls. The 1-point change in score from pre to post test is of clinical relevance.
change in signs and symptoms of major depression | baseline, 8 and 22 weeks later
  Cornell Scale for Depression in dementia (CSDD) contains 19 items evaluating signs and symptoms of major depression in individuals with dementia. Each item is rated for severity on a scale from 0 (absent) to 2 (severe). The information is collected through clinical observation and through two semi-structured interviews: one addressed to the caregiver and one to the person with dementia. The total score, given by the sum of the 19 items, if lower than 6 indicates the absence of depressive symptoms, if higher than 10 it indicates a probable major depression and finally if higher than 18 it indicates the presence of major depression
change in neuropsychiatric disturbances | baseline, 8 and 22 weeks later
  Neuropsychiatric Inventory (NPI) evaluates 12 neuropsychiatric disturbances common in dementia: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. A total NPI score and a total caregiver distress score are calculated. The total NPI score, which can range from 1 to 144, is the product of the frequency of manifestation and the severity of each disorder. Higher scores indicate more frequent and more severe behavioral problems

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pelliccioni, MD, Principal Investigator — IRCCS INRCA, Ancona, Italy
Locations (1):
- Cognitive Disorders and Dementia (CDCD) -INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gambella E, Margaritini A, Benadduci M, Rossi L, D'Ascoli P, Riccardi GR, Pasquini S, Civerchia P, Pelliccioni G, Bevilacqua R, Maranesi E. An integrated intervention of computerized cognitive training and physical exercise in virtual reality for people with Alzheimer's disease: The jDome study protocol. Front Neurol. 2022 Aug 12;13:964454. doi: 10.3389/fneur.2022.964454. eCollection 2022. PMID 36034306